CLINICAL TRIAL: NCT00838617
Title: Muscle Ultrasound: A New Tool for Measuring Progression in ALS
Brief Title: Muscle Ultrasound: A New Tool for Measuring Progression in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Christopher D. Lee, MD, Clinical Fellow, Department of Neurology, Vanderbilt University
Other Study IDs: 081243
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Ultrasonography; Atrophy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Participants with ALS: Participants diagnosed with ALS.

SUMMARY:
This is a study in patients with Amyotrophic Lateral Sclerosis (ALS). We will use muscle ultrasound as a tool to try and see if there are changes in muscle size that can find out how fast ALS is progressing. This might give us a better way to carry out further studies on new drugs to see if they might help slow the progression of ALS.

Participants in the study will have muscle ultrasound performed on a few muscles in the arms and legs at the first visit, and again 3 months later, and one last time 3 months after that. This takes about 10 minutes, is painless, and involves scanning the muscle with a handheld device, with some gel applied to the skin. At each visit, there will also be a questionnaire about symptoms and strength testing.

DETAILED DESCRIPTION:
Protocol for the Study - Muscle Ultrasound: A New Tool for Measuring Progression in ALS

A. Specific Aims The authors propose to study the change in muscle mass over time in patients with ALS. Muscle atrophy is a very common feature of the disease, and in clinical experience correlates with progressing weakness. As such, it is a qualitative marker of disease progress, although this lacks a quantitative marker. Muscle ultrasound is a safe, noninvasive, and rapid method of measuring muscle volume or thickness (1). Recently Arts, et al published an assessment of muscle ultrasound, specifically including reduced muscle depth and increased ultrasound echogenicity (2). We believe determining quantitatively the rate of progression of muscle mass in a group of patients with ALS will lead to a clinically useful tool to serve as a marker of disease progression, which may be useful in clinical trials for new therapies for this disease.

B. Background and Significance ALS is a quickly progressive disease that results in skeletal muscle weakness, including ventilatory weakness, which is the ultimate cause of death for the vast majority of patients with ALS. Median survival from diagnosis is less than 3 years. There is only one drug approved to treat ALS, riluzole, and its effects to limit the progression of the illness are slight (6). Current study designs often use a primary endpoint of either death from ALS or initiation of long-term mechanical ventilation (LTMV). There are other tools to assess progression, which can include a questionnaire called the ALS functional rating scale (ALS-FRS), a direct measurement of strength, or an electromyography technique called motor unit number estimate (MUNE). Each has potential drawbacks, which include potential lack of objectivity in questionnaire and variable effort when assessing direct strength measurements. There has also been work to correlate magnetic resonance spectroscopy findings to progression in ALS, with some positive results (3). However, this technology is expensive, time consuming, and not widely available. Muscle ultrasound may be sensitive enough to quantitatively detect changes in muscle thickness (4), which may serve as an objective tool to measure disease progression, for the purpose of clinical trials. Muscle echointensity (EI) is also abnormal in ALS (2, 4), although this assessment is less reliable among different observers and ultrasound settings, resulting in less diagnostic precision. Normal values for muscle thickness and echointensity are available, with norms varying by age and weight (5). Muscle ultrasound is readily available, noninvasive, inexpensive, and could be used in the context of a clinical examination. Muscle ultrasound is painless and can be completed in a few minutes.

C. Preliminary Studies/Progress Report As this is a pilot study, there is no preliminary data using muscle ultrasound longitudinally in patients with ALS. The study by Arts et al used muscle ultrasound to assist in the ALS diagnosis, but to our knowledge, muscle ultrasound has not been used to detect longitudinal changes in the illness. This study will help in the development of future studies testing pharmacologic agents in ALS, by providing muscle ultrasound as a validated endpoint in the progression of ALS.

D. Research Design and Methods Ten patients will be recruited to participate, and will have serial muscle ultrasound examinations every three months, at regularly scheduled clinic appointments in the Vanderbilt ALS clinic. Muscles examined will include forearm flexors, biceps, and tibialis anterior. The thickness of each muscle will be measured at standard sites for these muscles, in addition to the echogenicity as measured by a grayscale histogram representation. The rate of loss of ultrasound-measured muscle thickness will be assessed over time. Our hypothesis is that there will be significant loss of muscle thickness over time, which will correlate with disease severity. As different patients have different rates of deterioration, there will likely be significant differences in the rate of muscle volume loss from patient to patient. A secondary endpoint will be an increase over time in muscle echogenicity. Patients will complete the ALS Functional Rating Scale (ALSFRS-R), a 12 item subjective scale that assesses several motor functions, including function of speech, swallowing, respiration, and activities of daily living. Grip strength will be measured by hand grip dynamometry, using the best result from 3 attempts in each limb. Secondary analyses will also be conducted to correlate the decrease in ultrasound-measure muscle depth with the ALS Functional-Rating Scale, and with measures from hand grip dynamometry.

The study will be conducted over a period of 8 months. All patient data will be kept in a password-secured online database called REDcap. Any adverse events will be reported to the IRB, as none are expected with this safe diagnostic modality.

E. Inclusion Criteria

1. All patients must meet the El Escorial criterion for definite or probable ALS.
2. Patients forced vital capacity (FVC) must exceed 50%.

F. Exclusion Criteria

1. Patients with primary lateral sclerosis (PLS) and other forms of motor neuron disorders will not participate.
2. Patients with severe weakness from ALS who require continuous mechanical ventilation, who have a forced vital capacity less than 50%, or who have no clinically measurable strength in the arms and legs.
3. Patients without cognitive capacity to give informed consent. This is not a clinical feature of ALS, and therefore such patients would have an alternate diagnosis that would prevent such capacity.

G. Privacy/Confidentiality This is minimized by using study numbers, and labeling all patient data with study numbers and no other identifying information. The medical record numbers that correspond to each study number will be stored only in REDcap, a secure, password-protected database.

H. Human Subjects Research/Risks Careful consideration will be given to the protection of subjects from research risks and to the appropriate inclusion of women and minorities in the subjects who will be studied. Research risks are substantially limited by the noninvasive nature of muscle ultrasound, and the absence of any pharmacologic intervention in the study. There is a theoretical risk of breach of confidentiality, which is minimized as noted in the section above.

I. Reporting of Adverse Events/Unanticipated Problems involving Risk to Participants or Others The PI will report to the IRB in the event of an adverse event involving any participant, study personnel, or others, either from procedures involved in the study, or in the event of breach of participant confidentiality. These risks are minimized as noted above.

J. Statistical Considerations As this is a pilot study, this is not powered to likely find a statistically significant difference. Nonetheless, a mixed effect model statistical evaluation of the changes in muscle ultrasound values will be carried out for analysis.

K. Follow-up and Record Retention At the conclusion of the study, the study data will be maintained electronically only, in secure, encrypted format by the PI on REDcap for 6 years. After that time, any data not submitted to the patient's StarPanel electronic record will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* must meet the El Escorial criterion for definite or probable ALS.
* forced vital capacity (FVC) must exceed 50%.

Exclusion Criteria:

* Patients with primary lateral sclerosis (PLS) and other forms of motor neuron disorders
* severe weakness from ALS who require continuous mechanical ventilation, who have a forced vital capacity less than 50%, or who have no clinically measurable strength in the arms and legs.
* Patients without cognitive capacity to give informed consent. (This is not a clinical feature of ALS, and therefore such patients would have an alternate diagnosis that would prevent such capacity.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ALS (Amyotrophic Lateral Sclerosis)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Muscle thickness, as measured by muscle ultrasound, will decrease over time in patients with ALS. | 6 months

SECONDARY OUTCOMES:
Muscle thickness, as measured by muscle ultrasound, will correlate with decline in strength testing. | 6 months
Muscle thickness, as measured by muscle ultrasound, will correlate with decline in the ALS-FRS (ALS Functional Rating Scale) over time. | 6 months
Muscle echogenicity, as measured by muscle ultrasound, will increase in time, and will correlate with loss of muscle strength. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Lee, MD, Principal Investigator — Vanderbilt University Medical Center; Peter D Donofrio, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- ALS Clinic, Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Walker FO. Neuromuscular ultrasound. Neurol Clin. 2004 Aug;22(3):563-90, vi. doi: 10.1016/j.ncl.2004.03.004. PMID 15207876
- [Background] Arts IM, van Rooij FG, Overeem S, Pillen S, Janssen HM, Schelhaas HJ, Zwarts MJ. Quantitative muscle ultrasonography in amyotrophic lateral sclerosis. Ultrasound Med Biol. 2008 Mar;34(3):354-61. doi: 10.1016/j.ultrasmedbio.2007.08.013. Epub 2007 Oct 26. PMID 17964067
- [Background] Unrath A, Ludolph AC, Kassubek J. Brain metabolites in definite amyotrophic lateral sclerosis. A longitudinal proton magnetic resonance spectroscopy study. J Neurol. 2007 Aug;254(8):1099-106. doi: 10.1007/s00415-006-0495-2. Epub 2007 Apr 13. PMID 17431700
- [Background] Pillen S, Arts IM, Zwarts MJ. Muscle ultrasound in neuromuscular disorders. Muscle Nerve. 2008 Jun;37(6):679-93. doi: 10.1002/mus.21015. PMID 18506712
- [Background] Arts IM, Pillen S, Overeem S, Schelhaas HJ, Zwarts MJ. Rise and fall of skeletal muscle size over the entire life span. J Am Geriatr Soc. 2007 Jul;55(7):1150-2. doi: 10.1111/j.1532-5415.2007.01228.x. No abstract available. PMID 17608902
- [Background] Lacomblez L, Bensimon G, Leigh PN, Guillet P, Meininger V. Dose-ranging study of riluzole in amyotrophic lateral sclerosis. Amyotrophic Lateral Sclerosis/Riluzole Study Group II. Lancet. 1996 May 25;347(9013):1425-31. doi: 10.1016/s0140-6736(96)91680-3. PMID 8676624
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847